CLINICAL TRIAL: NCT04251819
Title: Buprenorphine Plus Baclofen to Increase Analgesia in Healthy Volunteers
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No funding for this project
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Cropsey, Professor of Psychiatry, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300004505
Record Dates: First submitted 2019-12-18; First posted 2020-02-05 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Acute Pain; Analgesia
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Baclofen

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants randomized to this arm will receive one dosage of Placebo as part of their second study appointment.
  Interventions: Drug: Placebos
- Baclofen 5mg (Experimental): Participants randomized to this arm will receive one dosage of 5 mg of Baclofen as part of their second study appointment.
  Interventions: Drug: Baclofen 5 mg
- Baclofen 10mg (Experimental): Participants randomized to this arm will receive one dosage of 10 mg of Baclofen as part of their second study appointment.
  Interventions: Drug: Baclofen 10mg

INTERVENTIONS:
Drug: Placebos — Participants will receive placebo in combination with 0.3 mg of buprenorphine to examine analgesia in acute pain tasks.
  Arms: Placebo
Drug: Baclofen 5 mg — Participants will receive 5mg of baclofen in combination with 0.3 mg of buprenorphine to examine analgesia in acute pain tasks.
  Arms: Baclofen 5mg
Drug: Baclofen 10mg — Participants will receive 10mg of baclofen in combination with 0.3 mg of buprenorphine to examine analgesia in acute pain tasks.
  Arms: Baclofen 10mg

SUMMARY:
To determine if baclofen will enhance buprenorphine analgesia for acute pain in healthy volunteers.

DETAILED DESCRIPTION:
Abuse of opioids is a significant and growing problem in the United States. In the past two decades, opioid prescriptions have quadrupled while the age of heroin initiation has decreased, suggesting that more individuals are using opioids and transitioning to heroin and potent synthetic opioids than in the past. Further, fatal opioid overdose is now the leading cause of accidental death and is the 5th highest overall cause of mortality in the US. Engaging opioid users in opioid agonist treatments has been shown to lower rates of criminal behavior, lower rates of non-opioid drug use, and increase retention in drug treatment programs, while decreasing mortality and new HIV and hepatitis infections. However, a recent study noted that 68% of patients prescribed buprenorphine had poor medication adherence, which was associated with illicit opioid use. A Cochrane review concluded that buprenorphine was less effective at retaining patients in treatment relative to methadone. One reason for lower treatment retention may be the high comorbidity of opioid use disorder and chronic pain and/or opioid-induced hyperalgesia. Buprenorphine, as a partial mu agonist, provides lower analgesia but an improved safety profile relative to full agonists like methadone. Thus, enhancing the analgesic properties of buprenorphine will provide a safer alternative for opioid use disorder patients with chronic pain/hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* general good health
* English speaking

Exclusion Criteria:

* Pregnant or nursing
* Opioid use disorder or any substance use disorder other than nicotine
* Prescribed agonist treatment for opioid dependence or prescribed opioids for a medical condition
* Prescribed naltrexone
* Known sensitivity to buprenorphine, naloxone, or baclofen
* Acute or chronic pain condition
* Trouble breathing or a pulmonary condition
* Prescribed benzodiazepines or daily use of benzodiazepines
* Positive drug screen (positive cannabis result allowed)
* Cognitive impairment or psychiatric disorder requiring treatment
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Cropsey, Psy.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants randomized to this arm will receive Placebo.
- Baclofen 5mg: Participants randomized to this arm will receive 5 mg of Baclofen.
- Baclofen 10mg: Participants randomized to this arm will receive 10 mg of Baclofen.
Period: Overall Study
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Started | 6 | 8 | 5
Completed | 6 | 8 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg | Total
Number analyzed (Participants) | 6 | 8 | 5 | 38
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 6 | 8 | 5 | 19
  (all) | 27.17 (12.58) | 36.63 (11.89) | 22.8 (2.59) | 29.58 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 6 | 8 | 5 | 19
  Female | 2 | 8 | 2 | 12
  Male | 4 | 0 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  number analyzed (Participants) | 6 | 8 | 5 | 19
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 5 | 4 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  number analyzed (Participants) | 6 | 8 | 5 | 19
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: number analyzed (Participants) | 6 | 8 | 5 | 19
  United States | 6 | 8 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pain Threshold
Description: Pain threshold refers to the intensity at which a stimulus is first perceived as painful. Heat stimuli will be delivered using a computer-controlled thermal stimulation system with a 30 millimeter X 30 millimeter probe. From a baseline of 32 degrees Celsius, the probe temperature will increase at a rate of .5 degrees Celsius/second until the participant responds by pressing a button on a handheld device. For heat pain threshold, participants will be instructed to press the button when the sensation "first becomes painful" Pain rating scores will be reflected in scores of 0-100, 0 being the least amount of pain and 100 being the most amount of pain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 8 | 5
Degrees Celsius | 44.62 (2.13) | 45.11 (3.04) | 43.56 (3.77)

2. Primary Outcome: Pain Threshold
Description: as for outcome 1
Time Frame: 1.5 hours post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 5 | 8 | 5
Degrees Celsius | 43.82 (2.46) | 43.95 (2.70) | 42.06 (3.14)

3. Primary Outcome: Pain Tolerance
Description: Pain tolerance refers to the maximum amount of pain produced by a stimulus that a person is able/willing to tolerate. Heat stimuli will again be delivered using the computer-controlled thermal stimulation system. From a baseline of 32 degrees Celsius, the probe temperature will increase at a rate of .5 degrees Celsius/second until the participant responds by pressing a button on a handheld device. For heat pain tolerance, participants will be instructed to press the button when they are "no longer willing to tolerate" the painful sensation. Pain rating scores will be reflected in scores of 0-100, 0 being the least amount of pain and 100 being the most amount of pain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 8 | 5
Degrees Celsius | 48.17 (1.52) | 46.84 (2.00) | 47.34 (2.11)

4. Primary Outcome: Pain Tolerance
Description: as for outcome 3
Time Frame: 1.5 hours post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 5 | 8 | 5
Degrees Celsius | 47.84 (1.86) | 47.70 (2.20) | 46.36 (2.56)

5. Primary Outcome: Temporal Summation of Pain
Description: Temporal summation of pain refers to a form of endogenous pain facilitation characterized by the perception of increased pain despite constant or even reduced peripheral afferent input. Temporal summation is presumed to be the psychophysical manifestation of wind-up. Wind-up is a phenomenon where repetitive stimulation of C primary afferents at rates greater than 0.3 Hertz produces a slowly increasing response of second-order neurons in the spinal cord. Pain rating scores will be reflected in scores of 0-100, 0 being the least amount of pain and 100 being the most amount of pain.
Time Frame: Baseline
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 5 | 5 | 4
units on a scale | 43.2 (8.0) | 48.4 (35.5) | 60.25 (35.3)

6. Primary Outcome: Temporal Summation of Pain
Description: as for outcome 5
Time Frame: 1.5 hours post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 5 | 6 | 3
units on a scale | 47.6 (17.5) | 64.5 (23.0) | 36.7 (23.6)

7. Primary Outcome: Conditioned Pain Modulation
Description: A routinely used quantitative sensory testing protocol for the measurement of endogenous pain inhibition is conditioned pain modulation, which refers to the reduction in pain from one stimulus (the test stimulus) produced by the application of a second pain stimulus at a remote body site (the conditioning stimulus). Conditioned pain modulation is believed to reflect the perceptual manifestation of diffuse noxious inhibitory controls, whereby ascending projections from one noxious stimulus activate supraspinal structures that trigger descending inhibitory projections to the dorsal horn. Pain rating scores for the test stimulus and the conditioning stimulus will be reflected in scores of 0-100, 0 being the least amount of pain and 100 being the most amount of pain. The conditioned pain modulation score is the difference between the two pain rating scores.
Time Frame: Baseline
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 7 | 5
units on a scale | -0.2 (7.4) | 2.1 (15.5) | -2.0 (5.7)

8. Primary Outcome: Conditioned Pain Modulation
Description: as for outcome 7
Time Frame: 1.5 hours post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 5 | 6 | 4
units on a scale | 3.0 (5.7) | -10.8 (15.0) | -6.3 (4.8)

9. Primary Outcome: Suprathreshold Pain Response
Description: Ratings of pain in response to discrete stimuli with intensities above the pain threshold detection/ patients provide an intensity rating using any number of a 0-100 scale whereby 0=no pain and 100= the most intense pain imaginable
Time Frame: Baseline
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 6 | 5
units on a scale | 42.5 (20.4) | 54.2 (34.7) | 53.4 (37.6)

10. Primary Outcome: Suprathreshold Pain Response
Description: as for outcome 9
Time Frame: 1.5 hours post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 5 | 8 | 5
units on a scale | 36.0 (15.2) | 68.8 (20.8) | 54.0 (30.7)

11. Secondary Outcome: Opioid Symptom Checklist
Description: Measures the amount and intensity of side effects after being administered an opioid. The measure consists of 14 questions about potential opioid symptoms, and each the severity of the symptom is rated on a scale from 0 to 4, with 0 reflecting not at all feeling or being bothered by the symptom and 4 reflecting being severely bothered by the symptom. The score is the sum of the 14 responses. The minimum value is 0 and the maximum value is 56.
Time Frame: 30 minutes post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 8 | 5
units on a scale | 4.67 (4.08) | 0.75 (1.39) | 0.60 (0.54)

12. Secondary Outcome: 26-item Visual Analog Scale (VAS)
Description: Measures subjective and physiological effects of a medication using mood states as well as questions about the dose of medication. The measure consists of 7 questions about potential drug effects, and each response is rated on a scale of 0 to 100, with 0 reflecting not at all feeling the effect and 100 reflecting very much feeling the effect. The score is the sum of the 7 responses. The minimum value is 0 and the maximum value is 700.
Time Frame: 30 minutes post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 8 | 5
units on a scale | 180.7 (94.3) | 50.4 (88.5) | 120.2 (76.9)

13. Secondary Outcome: Drug Effects Questionnaire-5
Description: Measures subjective experiences of a drug. The measure consists of 5 questions about the participant's experience of the drug effects, and each response is rated on a scale of 0 to 100, with 0 reflecting not at all having an experience and 100 reflecting extremely having that experience. The score is the sum of the 5 responses. The minimum value is 0 and the maximum value is 500.
Time Frame: 30 minutes post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Population: Data were missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 7 | 5
units on a scale | 168.8 (106.7) | 101.1 (76.0) | 103.8 (65.9)

14. Secondary Outcome: 26-item Visual Analog Scale ("Subjective Drug Effects")
Description: This 26-item VAS measures subjective and physiological effects of a medication using mood states as well as questions about the dose of medication. The measure consists of 7 questions about potential drug effects, and each response is rated on a scale of 0 to 100, with 0 reflecting not at all feeling the effect and 100 reflecting very much feeling the effect. The score is the sum of the 7 responses. The minimum value is 0 and the maximum value is 700.
Time Frame: 30 minutes post-drug administration during session 2, occurs 7 ± 2 days after baseline visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
Number analyzed (Participants) | 6 | 8 | 5
units on a scale | 180.7 (94.3) | 50.4 (88.5) | 120.2 (76.9)

ADVERSE EVENTS:
Time Frame: From baseline to 48 hours after dose session
Arm/Group | Placebo | Baclofen 5mg | Baclofen 10mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 0/8 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Baclofen 5mg (N=8) | Baclofen 10mg (N=5)
Emergency Department Visit (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Participant experienced nausea, dizziness, and vomiting shortly after receiving 4mg buprenorphine. Zofran did not relieve symptoms. Participant received saline IV and Zofran in the ED and was released the same day. No lingering effects the next day.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Baclofen 5mg (N=8) | Baclofen 10mg (N=5)
Buprenorphine Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Participant experienced dizziness, nausea, and vomiting after receiving 4mg buprenorphine. Participant reported grogginess and dizziness the next day, but nausea did not persist to the next day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT04251819/Prot_004.pdf
  • Statistical Analysis Plan (2025-11-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT04251819/SAP_007.pdf